CLINICAL TRIAL: NCT01235507
Title: Actemra - Local Bosnian Open, Multicentric, Trial to Evaluate Safety, Tolerability and Efficacy of Tocilizumab in Combination With Methotrexate in Patients With Active Rheumatoid Arthritis After Inadequate Response to DMARDs
Brief Title: A Study of RoActemra/Actemra (Tocilizumab) in Combination With Methotrexate in Patients With Active Rheumatoid Arthritis Who Have an Inadequate Response to Disease-Modifying Antirheumatic Drugs (DMARDs) (ALABASTER)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25303
Record Dates: First submitted 2010-10-15; First posted 2010-11-05 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; tocilizumab

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: methotrexate; Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: methotrexate — stable dose as prescribed
Drug: tocilizumab [RoActemra/Actemra] — 8 m/kg (maximum 800 mg) intravenously every 4 weeks for a total of 6 infusions

SUMMARY:
This open-label, single arm study will assess the safety and efficacy of RoActem ra/Actemra (tocilizumab) in combination with methotrexate in patients with activ e moderate to severe rheumatoid arthritis who have an inadequate response to dis ease-modifying antirheumatic drugs (DMARDs). Patients will receive RoActemra/Act emra at a dose of 8 mg/kg (maximum 800 mg) intravenously every 4 weeks for a tot al of 6 infusions. Methotrexate will be continued at a stable dose. Anticipated time on study treatment is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Active moderate to severe rheumatoid arthritis (RA)
* On methotrexate treatment (oral or parenteral) for at least 12 weeks, at stable dose of at least 15 mg/week for at least 6 weeks
* Oral corticosteroids must have been at stable dose of </= 10 mg/day prednisone (or equivalent) for at least 25 out of 28 days prior to first dose of study drug
* Body weight </= 150 kg

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months of study entry
* Rheumatic autoimmune disease other than RA
* Functional class IV according to American College of Rheumatology (ACR) classification
* Prior history of or current inflammatory joint disease other then RA
* Treatment with traditional DMARDs other than methotrexate within 1 month (for leflunomide 3 months) prior to baseline
* Treatment with any biologic drug that is used in the treatment or RA
* Intraarticular or parenteral corticosteroids within 6 weeks prior to baseline
* Known active current or history of recurrent infection
* History of or currently active primary or secondary immunodeficiency
* Positive for HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Bosnia and Herzegovina (3):
  - Banja Luka
  - Sarajevo
  - Tuzla

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab Plus Methotrexate (MTX): Participants received tocilizumab 8 milligrams per kilogram (mg/kg) (maximum 800 mg) intravenously (IV) every 4 weeks for a total of 6 infusions along with methotrexate stable dose as prescribed. Participants also received a stable dose of at least 5 mg per week (mg/week) of folate (or equivalent) given as either a single dose or divided into daily doses to achieve at least 5 mg/week, per investigator discretion.
Period: Overall Study
Arm/Group | Tocilizumab Plus Methotrexate (MTX)
Started | 71
Completed | 69
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: all participants enrolled in the study who completed the baseline visit and received at least 1 dose of study medication.
Groups:
- Tocilizumab Plus MTX: Participants received tocilizumab 8 mg/kg (maximum 800 mg) IV every 4 weeks for a total of 6 infusions along with methotrexate stable dose as prescribed. Participants also received a stable dose of at least 5 mg/week of folate (or equivalent) given as either a single dose or divided into daily doses to achieve at least 5 mg/week, per investigator discretion.
Arm/Group | Tocilizumab Plus MTX
Number analyzed (Participants) | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.76 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 10

OUTCOME MEASURES:

1. Secondary Outcome: Mean Disease Activity Score Based on 28 Joint Count (DAS28) by Visit
Description: DAS28 was calculated using the 28 joints count, the C-reactive protein levels (CRP) and participant's global assessment (PtGA) of disease activity. The following formula was used to determine DAS28.
  DAS28 (equals) = 0.56 × (square root of) √(TJC28) + 0.28 × √(SJC28) + 0.36 × ln(CRP+1) + 0.014 × GH + 0.96 where, TJC28 = tender joint count on 28 joints, SJC28 = swollen joint count on 28 joints, ln = natural log, CRP = C-reactive protein (mg/L), and GH = general health, determined by participant's global assessment of disease activity (100- millimeter [mm] visual analog scale [ VAS]).
  The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity.
Time Frame: Baseline, Weeks 8, 16 and 24
Population: ITT Population; number (n) = number of participants analyzed for the given parameter at the specified time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab Plus MTX
Number analyzed (Participants) | 71
units on a scale
  Baseline (n=71) | 6.28 (1.06)
  Week 8 (n=71) | 3.84 (1.29)
  Change from Baseline to Week 8 (n=71) | -2.44 (0.98)
  Week 16 (n=71) | 3.19 (1.23)
  Change from Baseline to Week 16 (n=71) | -3.09 (1.01)
  Week 24 (n=69) | 2.65 (1.23)
  Change from Baseline to Week 24 (n=69) | -3.62 (1.22)
Statistical Analysis 1: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 8; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 16; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test
Statistical Analysis 3: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 24; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test

2. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) and Clinical Remission (CR) as Assessed Using DAS28
Description: DAS28 was calculated using the 28 joints count, the CRP and PtGA of disease activity. The following formula was used to determine DAS28.
  DAS28 = 0.56 × √(TJC28) + 0.28 × √(SJC28) + 0.36 × ln(CRP+1) + 0.014 × GH + 0.96 where, TJC28 = tender joint count on 28 joints, SJC28 = swollen joint count on 28 joints, ln = natural log, CRP = C-reactive protein (mg/L), and GH = general health, determined by participant's global assessment of disease activity (100-mm VAS).
  The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. Participants were considered to have low disease activity when DAS28 was less than or equal to (≤) 3.2 and in clinical remission when DAS28 scores were less than (<) 2.6
Time Frame: Weeks 8, 16 and 24
Population: ITT Population; n= number of participants analyzed for the given parameter at the specified time point
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Plus MTX
Number analyzed (Participants) | 71
percentage of participants
  Week 8 CR (n=71) | 14.1
  Week 8 LDA (n=71) | 31.0
  Week 16 CR (n=71) | 39.4
  Week 16 LDA (n=71) | 49.3
  Week 24 CR (n=69) | 47.8
  Week 24 LDA (n=69) | 71.0

3. Secondary Outcome: Swollen and Tender Joint Counts
Description: 66 and 68 joints were assessed by the physician for tenderness or swelling respectively. The joints were counted as tender/not tender (tender=1; not tender=0) and swollen/not swollen (swollen=1; not swollen=0) and scored. The scores ranged from 0 to 66 for TJC and 0 to 68 for SJC. A negative change from baseline represents an improvement.
Time Frame: Baseline, Weeks 8, 16 and 24
Population: ITT Population; n= number of participants analyzed for the given parameter at the specified time point
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Tocilizumab Plus MTX
Number analyzed (Participants) | 71
Joints
  Baseline SJC (n=71) | 19.48 (10.97)
  Week 8 SJC (n=71) | 6.72 (5.76)
  Change in SJC from Baseline to Week 8 (n=71) | -12.76 (10.93)
  Week 16 SJC (n=71) | 3.73 (4.88)
  Change in SJC from Baseline to Week 16 (n=71) | -15.75 (9.59)
  Week 24 SJC (n=69) | 2.43 (4.12)
  Change in SJC from Baseline to Week 24 (n=69) | -16.83 (9.51)
  Baseline TJC (n=71) | 24.62 (11.84)
  Week 8 TJC (n=71) | 10.59 (8.38)
  Change in TJC from Baseline to Week 8 (n=71) | -14.03 (12.21)
  Week 16 TJC (n=71) | 7.12 (7.25)
  Change in TJC from Baseline to Week 16 (n=71) | -17.49 (11.02)
  Week 24 TJC (n=69) | 5.03 (5.97)
  Change in TJC from Baseline to Week 24 (n=69) | -19.48 (10.27)
Statistical Analysis 1: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 8; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 16; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test
Statistical Analysis 3: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 24; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test

4. Secondary Outcome: Physician's Global Assessment of Disease Activity
Description: Physician's global assessment of disease activity was performed using a 100 mm VAS ranging from no arthritis activity (0) to maximal arthritis activity (100). The distance in mm from the left edge of the scale was measured. Higher scores indicated higher disease activity. A negative change from baseline represents an improvement.
Time Frame: Baseline, Weeks 8, 16 and 24
Population: ITT Population; n=number of participants analyzed for the given parameter at the specified time point
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab Plus MTX
Number analyzed (Participants) | 71
mm
  Baseline (n=71) | 67.44 (17.72)
  Week 8 (n=71) | 35.99 (20.53)
  Change from Baseline to Week 8 (n=71) | -31.45 (17.76)
  Week 16 (n=71) | 26.48 (20.48)
  Change from Baseline to Week 16 (n=71) | -40.97 (20.7)
  Week 24 (n=69) | 19.28 (17.48)
  Change from Baseline to Week 24 (n=69) | -48.09 (19.69)
Statistical Analysis 1: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 8; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 16; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test
Statistical Analysis 3: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 24; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test

5. Secondary Outcome: Participant's Global Assessment of Disease Activity
Description: Participant's global assessment of disease activity was performed using a 100 mm VAS ranging from no arthritis activity (0) to maximal arthritis activity (100). The distance in mm from the left edge of the scale was measured. Higher scores indicated higher disease activity. A negative change from baseline represents an improvement.
Time Frame: Baseline, Weeks 8, 16 and 24
Population: ITT Population; n=number of participants analyzed for the given parameter at the specified time point
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab Plus MTX
Number analyzed (Participants) | 71
mm
  Baseline (n=71) | 70 (16.84)
  Week 8 (n=71) | 42.87 (20.67)
  Change from Baseline to Week 8 (n=71) | -27.13 (21.60)
  Week 16 (n=71) | 33.20 (21.16)
  Change from Baseline to Week 16 (n=71) | -36.80 (22.43)
  Week 24 (n=69) | 24.56 (20.15)
  Change from Baseline to Week 24 (n=69) | -45.30 (22.74)
Statistical Analysis 1: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 8; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 16; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test
Statistical Analysis 3: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 24; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test

6. Secondary Outcome: Participant's Global Assessment of Pain
Description: Participant's global assessment of pain was performed using a 100 mm VAS ranging from no pain (0) at the left edge to unbearable pain (100) at the right edge. The distance in mm from the left edge of the scale was measured. A negative change from baseline represents an improvement.
Time Frame: Baseline, Weeks 8, 16 and 24
Population: ITT Population; n=number of participants analyzed for the given parameter at the specified time point
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab Plus MTX
Number analyzed (Participants) | 71
mm
  Baseline (n=71) | 69.73 (17.60)
  Week 8 (n=71) | 42.34 (19.25)
  Change from Baseline to Week 8 (n=71) | -27.39 (19.44)
  Week 16 (n=71) | 33.94 (21.05)
  Change from Baseline to Week 16 (n=71) | -35.79 (21.52)
  Week 24 (n=69) | 25.54 (21.37)
  Change from Baseline to Week 24 (n=69) | -44.04 (25.11)
Statistical Analysis 1: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 8; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 16; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test
Statistical Analysis 3: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 24; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test

7. Secondary Outcome: CRP Levels
Description: CRP is a marker of acute phase inflammation and is measured in mg/L. A negative change from baseline represents an improvement.
Time Frame: Baseline, Weeks 8, 16 and 24
Population: ITT Population; n=number of participants analyzed for the given parameter at the specified time point
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Tocilizumab Plus MTX
Number analyzed (Participants) | 71
mg/L
  Baseline (n=62) | 11.98 (15.04)
  Week 8 (n=65) | 5.11 (14.12)
  Change from Baseline to Week 8 (n=61) | -6.68 (17.88)
  Week 16 (n=67) | 3.84 (11.91)
  Change from Baseline to Week 16 (n=60) | -8.0 (18.39)
  Week 24 (n=68) | 5.53 (14.07)
  Change from Baseline to Week 24 (n=60) | -5.97 (21.12)
Statistical Analysis 1: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 8; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 16; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test
Statistical Analysis 3: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 24; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test

8. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: ESR is a marker of inflammation and is measured in millimeters per hour (mm/hour). A negative change from baseline represents an improvement.
Time Frame: Baseline, Weeks 8, 16 and 24
Population: ITT Population; n=number of participants analyzed for the given parameter at the specified time point
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | Tocilizumab Plus MTX
Number analyzed (Participants) | 71
mm/hour
  Baseline (n=71) | 36.13 (24.82)
  Week 8 (n=71) | 9.04 (8.83)
  Change from Baseline to Week 8 (n=71 | -27.09 (22.98)
  Week 16 (n=71) | 8.71 (6.39)
  Change from Baseline to Week 16 (n=71) | -27.42 (23.07)
  Week 24 (n=69) | 10.3 (12.81)
  Change from Baseline to Week 24 (n=69) | -25.72 (27.54)
Statistical Analysis 1: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 8; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 16; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test
Statistical Analysis 3: Comparison: Tocilizumab Plus MTX; Change from Baseline to Week 24; Test type: Superiority or Other; p < 0.0005, Wilcoxon signed rank test

9. Primary Outcome: Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and AEs of Special Interest (AESIs)
Description: AEs, SAEs and AESI were recorded from the Screening Visit until the final visit at Week 24.
Time Frame: Screening Visit, Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: Safety Analysis Population: All participants enrolled in the study who received at least 1 dose of study medication and had at least 1 post-baseline assessment of safety (such as laboratory data, vital signs, or AEs) were included.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab Plus MTX
Number analyzed (Participants) | 71
percentage of participants
  AEs | 14.1
  SAE | 2.8
  AESI | 4.2

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the date of screening until the final visit at Week 24
Arm/Group | Tocilizumab Plus MTX
Serious Adverse Events (participants affected / at risk) | 2/71
Other Adverse Events (participants affected / at risk) | 7/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab Plus MTX (N=71)
Neoplasm - Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Exacerbation of RA (Immune system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab Plus MTX (N=71)
Leukocytopenia (Blood and lymphatic system disorders) | 3
Elevated AST (Hepatobiliary disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.